CLINICAL TRIAL: NCT01762995
Title: A Phase I, Open Label, Randomized, Four-Period Crossover Study to Evaluate the Effects of Calcium Carbonate 1200 mg and Ferrous Fumarate 324 mg on Pharmacokinetics of Dolutegravir 50 mg in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effects of Calcium Carbonate and Ferrous Fumarate on Pharmacokinetics of Dolutegravir in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 116898
Record Dates: First submitted 2012-12-19; First posted 2013-01-08 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-03

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: Dolutegravir, pharmacokinetics, calcium, iron, drug interaction, healthy volunteers
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir; Calcium Carbonate; ferrous fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Subjects in this cohort will take part in 4 treatment periods with one of the following treatments in each period. Subjects will receive all four treatments (one per period) in a random order. Treatment A = single dose DTG 50 mg fasted. Treatment B = single dose DTG 50 mg + Calcium Carbonate 1200 mg fasted. Treatment C = single dose of DTG 50 mg + Calcium Carbonate 1200 mg fed. Treatment D = single dose DTG 50 mg 2 hours prior to single dose Calcium Carbonate 1200 mg fasted
  Interventions: Drug: Dolutegravir 50 mg; Drug: Calcium Carbonate 1200 mg
- Cohort 2 (Experimental): Subjects in this cohort will take part in 4 treatment periods with one of the following treatments in each period. Subjects will receive all four treatments (one per period) in a random order. Treatment A = single dose DTG 50 mg fasted. Treatment E = single dose DTG 50 mg + Ferrous Fumarate 324 mg fasted. Treatment F = single dose of DTG 50 mg + Ferrous Fumarate 324 mg fed. Treatment G = single dose DTG 50 mg 2 hours prior to single dose Ferrous Fumarate 324 mg fasted
  Interventions: Drug: Dolutegravir 50 mg; Drug: Ferrous Fumarate 324 mg

INTERVENTIONS:
Drug: Dolutegravir 50 mg — One tablet ( 50 mg) will be administered orally as a single dose in each period per the random code
Drug: Calcium Carbonate 1200 mg — Two tablets (2 X 600 mg) will be administered orally as a single dose in three out of four periods to Cohort 1 only per the random code. Calcium carbonate will be given in fasted state, fed state and 2 hours before dolutegravir administration.
  Arms: Cohort 1
Drug: Ferrous Fumarate 324 mg — One tablet (324 mg) will be administered orally as a single dose in three out of four periods to Cohort 2 only per the random code. Ferrous fumarate will be given in fasted state, fed state and 2 hours before dolutegravir administration.
  Arms: Cohort 2

SUMMARY:
Human immune virus (HIV) infected subjects may take mineral supplements in combination with their antiretroviral medications. Calcium and Iron supplementations are commonly used and both of these have the potential to interact with Dolutegravir (DTG), this study will evaluate the potential of calcium and iron supplements to decrease DTG exposure. It will also evaluate two possible strategies for combined use; if an interaction is observed. The first strategy is a two hour separation. The second strategy involves the administration of DTG and the supplement with a meal since the presence of food modestly increases DTG exposure, and because mineral supplements can be administered with food.

This is an open label, randomized, two cohort, four-period cross-over study in healthy volunteers. One cohort will examine the effects of calcium carbonate and the other cohort will examine the effects of ferrous fumarate on the pharmacokinetic (PK) of DTG. Approximately 12 subjects will be enrolled into each of the two cohorts and receive each of four treatments in a randomized fashion: 1) A single dose of DTG 50 milligram (mg) administered under fasted conditions ; 2) A single dose of DTG 50 mg co-administered with a single dose of calcium carbonate or ferrous fumarate under fasted conditions ; 3) A single dose of DTG 50 mg co-administered with a single dose of calcium carbonate or ferrous fumarate with a moderate-fat meal; 4) A single dose of DTG 50 mg administered under fasted conditions 2 hours prior to administration of a single dose of calcium carbonate or ferrous fumarate. There will be a washout period of at least 7 days between treatments. Safety evaluations and serial PK samples will be collected during each treatment period. A follow-up visit will occur 7-14 days after the last dose of study drug. This study will be conducted at one center in the United States, with healthy adult male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECG.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: non-childbearing potential, or child-bearing potential and agrees to use one of the contraception methods for an appropriate period of time prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up visit.
* Body weight >= 50 kilogram (kg) for males and >=45 kg for females and body mass index (BMI) within the range 18.5 to 31.0 kg/meter^2 (inclusive).
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Single QT interval corrected using Fredericia's formula (QTcF) <450 millisecond (msec)
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive test for HIV antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine human chorionic gonadotropin test at screening or prior to dosing.
* Lactating females.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 gram of alcohol =12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GlaxoSmithKline (GSK) Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Unwillingness or inability to follow the procedures outlined in the protocol
* Subject is mentally or legally incapacitated.
* If heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* Consumption of red wine, Seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Unwillingness or inability to follow the procedures in the protocol.
* The subject's systolic blood pressure is outside the range of 90-140 millimeter mercury (mmHg, or diastolic blood pressure is outside the range of 45 to 90 mmHg or heart rate is outside the range of 50-100 beats per minutes (bpm) for female subjects or 45 to 100 bpm for male subjects. A single repeat is allowed for eligibility determination.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): Male subjects with Heart rate <45 and >110 bpm and female subjects with heart rate <50 and >100 bpm, PR <120 and >220 milliseconds (msec), QRS duration <70 and >120 msec, QTc (Bazett) >450 msec.
* Evidence of previous myocardial infarction (does not include ST segment changes associated with repolarization).
* Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome), non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats), and sinus pauses > 3 seconds.
* Any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety for the individual subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Single dose plasma DTG PK assessed by AUC (0-t) and AUC (0-infinity) | Blood samples (2 mililiter [mL]) for plasma PK parameters will be collected on Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hrs post-dose), Day 2 (24 and 36 hrs post-dose) and Day 3 (48 hrs post- dose) in each of the four treatment periods
  To evaluate the single dose PK of DTG, area under the concentration-time curve from time zero to last time of quantifiable concentration (AUC [0-t]) and area under the concentration-time curve from time zero extrapolated to infinite time (AUC (0-infinity) will be assessed with DTG given alone and when given with Calcium Carbonate (co-administered in fed or fasted state or 2 hours (hrs) separation, fasted) or Ferrous Fumarate (co-administered in fed or fasted state or 2 hrs separation, fasted)
Single dose plasma DTG PK assessed by Cmax and C24 | Blood samples (2 mL) for plasma PK parameters will be collected on Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hrs post-dose), day 2 (24 and 36 hrs post-dose) and day 3 (48 hrs post dose) in each of the four
  To evaluate the single dose PK of DTG, maximum observed concentration (Cmax) and concentration at 24 hours post-dose (C24) will be assessed with DTG given alone and when given with Calcium Carbonate (co-administered in fed or fasted state or 2 hrs separation, fasted) or Ferrous Fumarate (co-administered in fed or fasted state or 2 hrs separation, fasted)

SECONDARY OUTCOMES:
Safety and tolerability assessed by change from baseline in electrocardiogram (ECG) | Baseline and up to 36 days
  Single 12-lead ECGs will be obtained at each time point during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals.
Safety and tolerability assessed by number of subjects with adverse events (AEs) | up to 36 days
  AEs will be collected from the start of Study Treatment and until the follow-up contact
Safety and tolerability assessed by toxicity grading of clinical laboratory tests | up to 36 days
  Clinical laboratory tests include hematology, clinical chemistry, pregnancy test, alcohol and drug of abuse screen, and other additional parameters
Single dose plasma DTG PK assessed by AUC (0-24) | Blood samples (2 mL) for plasma PK parameter will be collected on day 1 (pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hrs post-dose), Day 2 (24 and 36 hrs post-dose) and Day 3 (48 hrs post- dose) in each of the four treatment periods.
  To evaluate the single dose PK of DTG, area under the concentration-time curve from time zero to 24 hrs post dose (AUC [0-24]) will be assessed when DTG will be given alone and when given with Calcium Carbonate (co-administered in fed or fasted state or 2 hrs separation, fasted) or Ferrous Fumarate (co-administered in fed or fasted state or 2 hrs separation, fasted)
Single dose plasma DTG PK assessed by tlag, tmax, and t1/2 | Blood samples (2 mL) for plasma PK parameter will be collected on Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hrs post-dose), Day 2 (24 and 36 hrs post-dose) and Day 3 (48 hrs post- dose) in each of the four treatment periods.
  To evaluate the single dose PK of DTG, lag time before observation of drug concentrations in sampled matrix (tlag), time of occurrence of Cmax (tmax), and terminal phase half-life (t1/2) will be assessed when DTG will be given alone and when given with Calcium Carbonate (co-administered in fed or fasted state or 2 hrs separation, fasted) or Ferrous Fumarate (co-administered in fed or fasted state or 2 hrs separation, fasted).
Single dose plasma DTG PK assessed by CL/F | Blood samples (2 mL) for plasma PK parameter will be collected on Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hrs post-dose), Day 2 (24 and 36 hrs post-dose) and Day 3 (48 hrs post- dose) in each of the four treatment periods.
  To evaluate the single dose PK of DTG, apparent clearance following oral dosing (CL/F) will be assessed when DTG will be given alone and when given with Calcium Carbonate (co-administered in fed or fasted state or 2 hrs separation, fasted) or Ferrous Fumarate (co-administered in fed or fasted state or 2 hrs separation, fasted).
Safety and tolerability assessed by change from baseline in blood pressure | Baseline and up to 36 days
  Blood pressure (BP) measurement will include systolic and diastolic BP measurement. BP will be measured after resting in a semi-supine position for 5 minutes
Safety and tolerability assessed by change from baseline in Pulse rate | Baseline and up to 36 days
  Pulse rate will be measured after resting in a semi-supine position for 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare